CLINICAL TRIAL: NCT01183286
Title: CFfone: A Cell Phone Support Program for Adolescents With Cystic Fibrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dawkins Productions, Inc. (Other)
Collaborators: University of Miami (Other); Columbia University (Other); University of Tennessee (Other); Children's National Research Institute (Other)
Responsible Party: Kevin Dawkins, Principal Investigator, Dawkins Productions, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 5R44HL088826-03 (NIH)
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CFFONE (Active Comparator)
  Interventions: Behavioral: CFFONE
- CF website (Placebo Comparator)
  Interventions: Behavioral: CF website

INTERVENTIONS:
Behavioral: CFFONE — A password-protected, secure website, which can be accessed via a web capable cell phone. The website contains age appropriate medical and behavioral information, disease management tools and social networking features for adolescents and young people who have Cystic Fibrosis.
  Arms: CFFONE
Behavioral: CF website — A CF-related educational website which has some areas of CF information and services relevant to adolescents.
  Arms: CF website

SUMMARY:
Adolescents with cystic fibrosis are particularly vulnerable to poor adherence, which negatively impacts their health status, quality of life and long term survival. CFFONE: A Cell Phone Support Program for Adolescents with Cystic Fibrosis, will make use of cutting-edge technology- a broadband capable, cellular telephone keyed into a highly-interactive informational web site. This web site will provide engaging online learning activities and resources specific to adolescents with cystic fibrosis. We believe the information and activities contained in CFFONE will improve adolescents knowledge, attitudes, and practices around cystic fibrosis and that adolescents exposed to the CFFONE program will demonstrate an increase in adherence to their treatment regimens and related improvements in their health status and quality of life.

DETAILED DESCRIPTION:
Generations of patients with cystic fibrosis (CF) have spent their childhoods fighting for breath and losing. Until recently, CF patients succumbed to this fatal, inherited lung disease as infants, young children or adolescents. With cutting-edge research spurring medical advances, each decade has shown improved survival, from a median life expectancy of 5 years in 1960, to 16 years in 1970, to 35 years today. Yet, the disease remains complex and adolescents with CF experience challenges that can reduce their adherence to treatment regimens and undermine their long-term well-being.

Poor adherence to complicated life long treatments impacts a patient's health and burdens the medical system. Adolescents are particularly vulnerable to poor adherence and its high costs. Even adolescents who experience comparatively mild symptoms of CF must follow a 3-hour treatment regimen every day, and medical experts report that their adherence ranges from poor (50% doing less than prescribed airway clearance regimen) to very poor (30% not doing any prescribed treatments).

CF can cause a host of social-emotional stressors, including uncertainty about the future, poor self-image, low self-esteem, and frustration with delayed growth/maturation all of which can impede adherence. Absences from school, being teased, keeping their illness secret, and lack of access to peers with CF due to risk of infection leave many adolescents with CF feeling isolated and alone. Due to parent over-protection and medical services that focus on symptoms, these patients often lack supportive coaching on issues (e.g., alcohol-and tobacco-related risks, sexual health, infection control, pain control, career prospects) that can impact the quality of their life.

This Phase II Randomized Control Trial (study) will test the hypothesis that adolescents with cystic fibrosis (CF) ages 11-17 (adolescent participants) and young adults with CF, ages 18-20 (adult participants) who access a password-protected, secure mobile website (CFFONE), via a web capable cell phone and use the site's age appropriate medical and behavioral information, disease management tools and social networking features will demonstrate: (1) an increase in CF knowledge- the primary end point of the study; (2) improved treatment adherence and improved quality of life- the secondary end points of the study and; (3) enhanced social support- the exploratory end point of the study, when compared to control group adolescent participants and adult participants.

To test this hypothesis, a longitudinal experimental design will be carried out in which participants will be randomly assigned to one of two conditions: cell phone access to CFFONE; or registering with a CF-related educational website containing CF information and services relevant to adolescents.

A recent National Institutes for Health solicitation for research to improve self-management and quality of life in children and adolescents with chronic diseases stated that, "Children with a chronic disease face a lifetime of careful health management requirements and lifestyle adaptations to prevent or manage related health complications. Interventions that make a difference in childhood disease self-management may set the stage for health outcomes later in life." (2003) We believe that CFFONE, with its innovative approach for enhancing self-management, has the potential to make that kind of difference in the lives of adolescents with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Cystic Fibrosis
* Be within the target age range of 11-20 years old at enrollment -Have regular access to an internet connected computer that does not prevent access to websites (i.e. a firewall) -

Exclusion Criteria:

-Have a developmental disorder that would affect ability to respond to survey questions -

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 146 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Cystic Fibrosis Knowledge Questionnaire (CFK) | The CFK will be administered at baseline, month 3, month 6 and month 9.
  The CFK assess participants' CF-related knowledge. The CFK consists of 42 multiple-choice items, with scores reported as percentage correct.

SECONDARY OUTCOMES:
Cystic Fibrosis Questionnaire-Revised (CFQ-R) | The CFQ-R will be administered at baseline, month 3, month 6 and month 9.
  To assess participants' quality of life the CFQ-R will be taken to measure the impact of CF on the participant's social functioning, respiratory symptoms and treatment burden. These three domains consist of 13 items. The adolescent/adult version will be used for participants 15-20 and the CFQ-R Older Child version will be used for participants ages 11-14.
Pharmacy Refill Data | Pharmacy Refill Data will be collected at baseline for the 12 months prior to enrollment; and again after the 9 month clinic visit for the 9 months of the study. The Prescribed Treatment Plan will be collected at baseline, month 3, month 6 and month 9.
  To measure treatment adherence a print out of CF related medications and refill data will be collected from participants' pharmacies. To obtain participant's prescription information in order to have adherence calculations for three month periods, the attending physician will fill out a prescribed treatment plan at every clinic visit during the study